CLINICAL TRIAL: NCT02986386
Title: Oral Health for Healthy Cognitive Aging
Acronym: SOECS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Pablo Galindo-Moreno, Professor, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SOECS-905
Record Dates: First submitted 2016-11-23; First posted 2016-12-08 (Estimated); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Malocclusion; Dementia
Keywords: Dental Occlusion; Oral Health; Mastication; Dementia; Psychological health
MeSH Terms: conditions — Malocclusion; Dementia; Bites and Stings; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Intervention 1 (Experimental): Dental occlusion restoration by placement of dental implants and prosthesis on missing teeth.
  Interventions: Procedure: Dental occlusion restoration
- Wait list control 1 (Other): Group of patients that will be evaluated until they receive the dental occlusion restoration procedure.
  Interventions: Procedure: Dental occlusion restoration
- Intervention 2 (Experimental): Orthodontic treatment of malocclusion.
  Interventions: Procedure: Orthodontic treatment of malocclusion
- Wait list control 2 (Other): Group of patients that will be evaluated until they receive the orthodontic treatment of malocclusion.
  Interventions: Procedure: Orthodontic treatment of malocclusion

INTERVENTIONS:
Procedure: Dental occlusion restoration — Placement of dental implants by surgical intervention followed, after a healing period of 2 months, by fabrication and installation of implant supported dental prosthesis
  Arms: Intervention 1; Wait list control 1
Procedure: Orthodontic treatment of malocclusion — Orthodontic therapy to treat malocclusion
  Arms: Intervention 2; Wait list control 2

SUMMARY:
Oral health is a critical factor of systemic health, although usually forgotten. A potential relation between cognitive deficits and oral diseases has been suggested. Adult cognitive dysfunctions have a high impact, not only economic, but social and in the family environment. Based on anatomical connectivity between the oral cavity and the central nervous system, the proposed study hypothesizes that masticatory function is a relevant determinant of human cognitive health. The restoration of canonical masticatory function and masticatory training could help to delay the development of such conditions. This project will also test if restoring phasic masticatory function improves the execution of cognitive tasks.

DETAILED DESCRIPTION:
Objective 1: To determine volumetric and anatomical changes of subcortical structures and cortical areas involved in the masticatory circuit and superior cognitive functions.

Objective 2: To determine the functional and brain connectivity changes associated with malocclusion and oral health.

Objective 3: To correlate the anatomic and functional changes associated with malocclusion and oral health with the performance of cognitive tasks representative of those executed in daily life.

ELIGIBILITY:
Inclusion Criteria:

* For Dental occlusion restoration groups: Need of, at least, two molar teeth replacement in the same quadrant.
* For Orthodontic treatment of malocclusion groups: Class I, II or III malocclusion.

Exclusion Criteria:

* Psychoactive drug.
* Central nervous system depressor.
* Patients not willing or not able to consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2016-11; Primary Completion 2023-01 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change of occlusion units | Baseline, 6, 12 and 36 months
  Number of teeth occluding with opposing teeth
Change of cerebral activity | Baseline, 6, 12 and 36 months
  Functional MRI
Change of cognitive function | Baseline, 6, 12 and 36 months
  Verbal fluency
Change of frame of mind | Baseline, 6, 12 and 36 months
  Beck test
Change of resting brain activity | Baseline, 6, 12 and 36 months
  Electroencephalographic activity

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Galindo-Moreno, DDS, PhD, Principal Investigator — Universidad de Granada
Locations (1):
- Facultad de Odontología, Granada, Spain

REFERENCES:
- [Background] Akazawa Y, Kitamura T, Fujihara Y, Yoshimura Y, Mitome M, Hasegawa T. Forced mastication increases survival of adult neural stem cells in the hippocampal dentate gyrus. Int J Mol Med. 2013 Feb;31(2):307-14. doi: 10.3892/ijmm.2012.1217. Epub 2012 Dec 18. PMID 23254518
- [Background] Elsig F, Schimmel M, Duvernay E, Giannelli SV, Graf CE, Carlier S, Herrmann FR, Michel JP, Gold G, Zekry D, Muller F. Tooth loss, chewing efficiency and cognitive impairment in geriatric patients. Gerodontology. 2015 Jun;32(2):149-56. doi: 10.1111/ger.12079. Epub 2013 Oct 16. PMID 24128078
- [Background] Gil-Montoya JA, Ponce G, Sanchez Lara I, Barrios R, Llodra JC, Bravo M. Association of the oral health impact profile with malnutrition risk in Spanish elders. Arch Gerontol Geriatr. 2013 Nov-Dec;57(3):398-402. doi: 10.1016/j.archger.2013.05.002. Epub 2013 Jun 10. PMID 23763956